CLINICAL TRIAL: NCT04323423
Title: Determining the Optimal Reduction in Sedentary Behaviour to Reduce Glycemic Variability and Maintain Cognition: a Randomized Control Trial
Brief Title: The DURATION Study: reDUcing sedentaRy behAviour to Maintain cogniTIve functiON.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator moved to a different role
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Professor, Western University, Canada
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Glycemic variability & SB
Record Dates: First submitted 2020-03-09; First posted 2020-03-26 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Sedentary Behavior; Mild Cognitive Impairment; Glucose Intolerance; Overweight and Obesity
Keywords: Sedentary Behaviour; Physical activity; Walking; Older adults; Cognition; Glycemic variability; Randomized controlled trial
MeSH Terms: conditions — Sedentary Behavior; Cognitive Dysfunction; Glucose Intolerance; Overweight; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized crossover trial and reported in accordance with CONSORT guidelines. The study will involve a total of three seven-day conditions (2 experimental and 1 control) with a three-week washout period in-between to minimize practice effects for a total intervention period of nine weeks. Each condition will consist of one day supervised in the laboratory followed by six at-home days, following lab protocol as closely as possible.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (CON) (No Intervention): 1) Condition A (CON): This will be the control condition. It will consist of uninterrupted sitting from 8 am until 7 pm, only rising from the chair to void.
- one 10 minute bout - (LONG) (Experimental): will consist of completing one 10-minute bout of light intensity walking (RPE 6-9) 30 minutes post-prandial. Participants will rise from their seated position to walk ~10 metres to a treadmill to perform this bout. The participant will repeat this after lunch and dinner, for an accumulated total of 30 minutes of light walking.
  Interventions: Behavioral: interrupting sedentary behaviour with light physical activity
- four 2.5 minute bouts SHORT (Experimental): will consist of interrupting sitting with four 2.5-minute bouts of light walking at 30 minutes, 60 minutes, 90 minutes and 120 minutes post-prandial. Participants will rise from their seated position to walk ~10 metres to a treadmill to perform these bouts. The participant will repeat this after breakfast, lunch and dinner for an accumulated total of 30 minutes of light walking.
  Interventions: Behavioral: interrupting sedentary behaviour with light physical activity

INTERVENTIONS:
Behavioral: interrupting sedentary behaviour with light physical activity — replacing sitting with light walking bouts at different frequencies/durations
  Arms: four 2.5 minute bouts SHORT; one 10 minute bout - (LONG)

SUMMARY:
Rationale: Older adults spend the majority of their time in sedentary behaviours (SB). High amounts of SB have been correlated with reduced cognitive performance. Long periods of time spent sitting results in excessive glycemic variability, potentially contributing to cognitive decline. Reducing/replacing SB with short intermittent bouts of light physical activity have shown positive effects on glycemic variability. Thus, interrupting prolonged sitting with bouts of light physical activity may regulate blood glucose and thus mitigate cognitive decline.

Purpose: This study intends to investigate the appropriate interval frequency of post-prandial SB reduction, by light physical activity needed to optimize total and incremental area under the curve for glucose response in overweight older adults at risk for glucose intolerance with mild cognitive impairment in both lab and free-living environments. Second, this study aims to investigate the acute impact of reducing SB on glycemic variability and its relationship with cognition.

Hypothesis: First, there will be a dose-dependent response of more frequent interruptions of SB (more frequent intervals of light physical activity) with better glycemic control. Second, reducing SB will result in less glycemic variability, which will translate into better levels of cognitive performance.

Methods: Generalized linear mixed models with random intercepts will be used to evaluate the differential effects of the experimental conditions on the selected outcomes.

DETAILED DESCRIPTION:
This study will be a randomized crossover trial and reported in accordance with CONSORT guidelines. The study will involve a total of three seven-day conditions (2 experimental and 1 control) with a three-week washout period in-between to minimize practice effects for a total intervention period of nine weeks (see figure 1). Each condition will consist of one day supervised in the laboratory followed by six at-home days, following lab protocol as closely as possible.

Participants will be referred to the study by their physician. Interested participants will be asked to contact the researcher by email or phone call. Interested Participants will be invited into the lab for a familiarization session. They will be instructed to avoid caffeine, alcohol and MVPA for 48 hours prior to this session. During this session the following information will be obtained;

* Written informed consent
* Height using a stadiometer and weight using a standard beam scale
* Demographics questionnaire (education, ethnicity, family background, comorbidities)
* Physical Activity Readiness Questionnaire (PARQ+) (Bredin, Gledhill, Jamnik, & Warburton, 2013)
* Resting blood pressure- will be measured once on each arm and then twice on the left arm with an automated BP monitor The participants will be educated/familiarized on the following;
* Cognitive assessments - Cambridge Neuropsychological Test Automated Battery (CANTAB)
* Fitting with an inclinometer (activPAL4)

Participants will be visited at their home ~72hrs prior to each condition to be fitted with the CGM and ActivPal. They will also be instructed to avoid caffeine, alcohol and MVPA for 48 hours prior to each of the three conditions. Dinner will be consumed between 7:00 and 9:00 pm, allowing for a 10 hour fast prior to the experimental condition the next morning. All participants will be instructed to arrive at the laboratory (with minimal activity during commute) at approximately 7:00 am. Upon arrival, participants will be asked to use the washroom and then rest for 30 minutes preceding a blood pressure measurement and first cognitive assessment. The participants will undergo the CANTAB cognitive assessments (at ~7:30 am) before meal consumption. A standardized breakfast meal will be consumed at 8:00 am, followed by lunch at 12:00 pm and dinner at 5:00 pm. Participants will be allotted 20 minutes for full meal consumption. The CANTAB cognitive assessments will then be re-administered at approximately 7:30 pm. Participants will be supervised throughout the conditions to ensure adherence to the protocols and will be permitted to watch DVDs, read books, magazines, newspapers, talk and/or work on a laptop computer. However, what they do during the first condition will be documented and then replicated for the remaining experimental conditions. Intensity of the bout intervals will be kept to an RPE of 6-9 using the Borg RPE scale.

Once the 12- hour laboratory component is complete, participants will be sent home (still wearing the CGM and activPAL) with the intension of replicating the laboratory-based protocol after each meal in their own free-living environment. Participants will track their mealtimes by sending photos to the researcher before consumption during the 6 at home days. The researcher will then go to the participants house on the last day (day 7) of each condition to re-administer the CANTAB cognitive assessments and collect the CGM, and activPal. There will then be a 3-week washout period, followed by replication of protocol for the remaining two conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Have a caregiver that works with you at least 20 hours a week (needs to be present for the familiarization session (explained below) and drop-off and pick-up from lab sessions)
* Diagnosis of diabetes by a healthcare provider (e.g. family doctor).
* Diagnosis of MCI by a healthcare provider
* Self-report being physically inactive (not meeting the current PA guidelines of 150 min MVPA/week)
* Self-report being sedentary- (defined as self-reported sedentary time ≥ 7 h/day)
* Able to walk one block without an assistive device
* Own a smartphone with unlimited outgoing text messages and access to internet connection. The smartphone must be either iphone 7 (with iOS of 12.2 or higher) or Android operating system 5 or higher to allow for Libre View mobile application compatibility.
* Able to read, write and understand English

Exclusion Criteria:

* Currently smoke
* Depression (Geriatric Depression Score short-form > 6 (GDS)) (Yesavage, Brink, Rose, & et al, 1983).
* Medication: hypoglycemics; antilipidemics; antidepressants; beta blockers; anti-anxiety agents
* Peri-menopausal or menopausal women (must be post-menopausal)
* Excessive alcohol consumption (> 8 points on the Alcohol Use Disorders Identification Test)
* Uncontrolled hypertension (measured systolic > 140 mmHg or diastolic > 90 mmHg)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Glycemic Variability | 1-7 days
  to investigate the appropriate interval frequency of post-prandial SB reduction, by light physical activity needed to optimize total and incremental area under the curve for glucose response in overweight older adults at risk for glucose intolerance with mild cognitive impairment in both lab and free-living environments.

SECONDARY OUTCOMES:
Cognition | 1-7 days
  CANTAB will be used to measure change in cognitive function. This is a computerized battery of neuropsychological tests utilizing touch sensitive screen technology that has been shown to be highly sensitive and a precise measure of cognitive function, correlated to neural networks (CANTAB, 2017). The following three cognitive domains were selected for testing; attention and psychomotor function (Motor Screening Task (MOT) and Rapid Visual Information Processing (RVP)), memory (Delayed Matching to Sample (DMS)) and executive function (Intra-Extra Dimensional Set Shift (IED))

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, Ph.D, Principal Investigator — Western University
Locations (1):
- The University of Western Ontario, London, Ontario, Canada